CLINICAL TRIAL: NCT06957574
Title: Erector Spinae Plane Block as Analgesia in Patients for Colectomy: A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block as Analgesia in Patients for Colectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Assistant professor, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESPB
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Colo-rectal Cancer
Keywords: erector spinae plane; colectomy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB (Active Comparator): ESPB using local anaesthetic 20 ml 0.25% bupivacaine on each side
  Interventions: Drug: Bubpivacaine
- Saline (Placebo Comparator): ESPB using normal saline 20 ml on each side
  Interventions: Drug: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Bubpivacaine — ESPB using local anesthetic 20 ml 0.25% bupivacaine on each side
  Arms: ESPB
Drug: Normal Saline (Placebo) — ESPB using normal saline 20 ml 0.25% bupivacaine on each side
  Arms: Saline

SUMMARY:
Management of postoperative pain relief is largely inadequate. Despite the recent advances in pain management, postoperative pain incidence has not decreased; most patients still experience severe pain after major surgery. Poorly or inadequately controlled pain was reported to be linked to prolonged hospitalization, decreased patient satisfaction, the risk of readmission, and a higher incidence of postoperative complications.

DETAILED DESCRIPTION:
In major abdominal surgeries, the gold standard for postoperative analgesia is thoracic epidural analgesia. Nevertheless, there are many concerns regarding its side effects, including motor blockade and hypotension. Moreover, many researchers interrogated its role as it may increase the risk of serious problems such as epidural hematoma and abscess. As an alternative, some surgeons proposed the transversus abdominis plane (TAP); however, a recent meta-analysis established that TAP block was of minimal effect.

The erector spinae plane block (ESPB) is a fairly original paraspinal plane block that was first designated for thoracic analgesia. Recently, some reports showed that it could offer effective and widespread somatic and visceral abdominal analgesia. Bilateral continuous ESP blockade represents a respected alternative to thoracic epidural analgesia. The local injection under the erector spinae muscle is carried out in this technique, which is estimated to spread a paravertebral of three vertebral levels cranially and four levels caudally. It was designated that the injected local anesthesia passes across the costotransverse foramina and blocks the ventral and dorsal rami of spinal nerves, causing a sensory blockade over the anterolateral thorax. The dermatomes enclosed by ESPB depend on the site of entry, the volume, and the concentration of the local anesthetic used. This RCT aimed to assess the analgesic effectiveness of US-guided bilateral erector spinae plane block in patients undergoing elective colectomy.

This randomized controlled trial was designed to assess the analgesic effectiveness of bilateral US-guided erector spinae plane blocks (ESPB) in patients undergoing elective colectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients of colorectal carcinoma scheduled for elective colectomy

Exclusion Criteria:

* Patients with a body mass index (BMI) of 35 kg/m2 or above
* patients with a history of hepatic or renal diseases
* patients with second- or third-degree heart blocks
* patients with coagulopathies
* patients with history of hypersensitivity to local anesthetics

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
morphine consumption | From the time of end of surgery till the pass of the first 24 hours postoperatively
  postoperative total morphine consumption over 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No